CLINICAL TRIAL: NCT02386085
Title: Patient-reported Adverse Events From Osteopathic Manipulative Treatment
Status: Completed | Type: Observational
Sponsor: A.T. Still University of Health Sciences (Other)
Collaborators: American Academy of Osteopathy (Other); A.T. Still Research Institute (Other Government); DO-Touch.NET (Unknown)
Responsible Party: Sponsor
Other Study IDs: OMT Adverse Events Study
Record Dates: First submitted 2015-03-06; First posted 2015-03-11 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Osteopathic Manipulative Treatment
Keywords: Osteopathic Manipulative Medicine; Osteopathic Manipulation; adverse effects; side effects; undesirable effects
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Osteopathic manipulative treatment (OMT): All participants will have received OMT to be eligible and will be followed for 1 week after treatment.
  Interventions: Procedure: Osteopathic manipulative treatment (OMT)

INTERVENTIONS:
Procedure: Osteopathic manipulative treatment (OMT) — OMT will be provided as part of the patient's health care, prior to enrollment in the study. All participants would have received the same intervention (OMT) if they had not enrolled in the study.

SUMMARY:
Currently, there is a significant deficiency in evidence regarding the safety of osteopathic manipulative treatments (OMT). To address this deficit, this study is designed to systematically evaluate the incidence and severity of OMT adverse events and examine the relationship of these adverse events to the technique(s) used and the body region(s) treated. The study is being conducted at the clinics of participating members of DO-Touch.NET, the only known practice-based research network (PBRN) focused on osteopathic manual medicine research. Eligible patients who receive OMT at one of the participating clinics will be asked to complete either a paper or online survey regarding any adverse events they experience within 1, 3, and 7 days following their treatment. Information regarding their diagnoses, which osteopathic techniques were used in their OMT, and which body regions were treated will be obtained from participant medical records. This data will be used to answer the following research questions:

1. What is the incidence of adverse events from osteopathic manipulative treatment?
2. What types of adverse events occur following osteopathic manipulative treatment?
3. Are there individual osteopathic techniques in particular body regions that have higher incidences of adverse events than other techniques or body regions?
4. Is the incidence of adverse events higher for some patient conditions than others?

ELIGIBILITY:
Inclusion Criteria:

* received osteopathic manipulative treatment at one of participating clinics

Exclusion Criteria:

* unable to communicate in English, Spanish, French, German, or Portuguese

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients who receive osteopathic manipulative treatment from a licensed practitioner for any reason.
Sampling Method: Non-Probability Sample
Enrollment: 1303 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Severity of adverse events related to osteopathic manipulative treatment (OMT) | Within 1 week after receiving OMT
  Data from surveys completed 24 hours, 72 hours, and 1 week after receiving OMT will be used to determine the severity, duration, and onset of symptoms/complaints experienced by participants. The 24- and 72-hour surveys assess the patient-reported severity, duration, and location of potential adverse events, as well as the existence and severity of these symptoms within the week prior to treatment and the participant's assessment of whether the symptom/complaint was related to the OMT they received. The 1-week survey will follow-up on symptoms/complaints reported on the 72-hour survey and whether participants have sought follow-up or urgent care, visited the emergency room, or been hospitalized during the week following OMT.

CONTACTS AND LOCATIONS:
Overall Officials: Jane C Johnson, MA, Principal Investigator — A.T. Still University of Health Sciences; Brian F Degenhardt, DO, Principal Investigator — A.T. Still University of Health Sciences

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-07-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT02386085/Prot_SAP_000.pdf
  • Informed Consent Form (2015-02-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT02386085/ICF_001.pdf